CLINICAL TRIAL: NCT04836468
Title: Changes in Blood Flow in the Lower Limb With the Application of Magnetic Tape in Patients With Low Back Pain. Double-blinded Clinical Trial.
Brief Title: Changes in Blood Flow in the Application of Magnetic Tape in Patients With Low Back Pain. RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Selva (Other)
Responsible Party: Sponsor-Investigator, Francisco Selva, PhD physiotherapy, Clínica Dr. Francisco Selva
Organization: Clínica Dr. Francisco Selva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
Keywords: magnetic tape; Pressure; Pain; Vascular; Ultrasound
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Application of Magnetic Tape transversely over the vertebral levels of L4 and L5
  Interventions: Diagnostic Test: Tape application
- Placebo group (Placebo Comparator): Application of kinesiology tape transversely over the vertebral levels of L4 and L5
  Interventions: Diagnostic Test: Tape application

INTERVENTIONS:
Diagnostic Test: Tape application — Magnetic Tape or Kinesiology tape will be applied randomly with both the examiner and the subjects blinded.

SUMMARY:
A tape is applied over the lumbar 4th and lumbar 5th levels crosswise in people with low back pain. The possible variation of the arterial flow of the femoral artery is measured with ultrasound. A kinesiology tape was used as placebo tape and Magnetic Tape was used as experimental randomly.

DETAILED DESCRIPTION:
A double-blind randomized clinical trial is designed where subjects with low back pain will be selected and blinded to recieve the Magnetic Tape® (tape with magnetic effects of less than 2 Gauss) or placebo Tape. Likewise, the evaluator who puts the Magnetic Tape® does not know what material he is using, as it is supplied by another researcher. The sonographer also does not know if the patient has low back pain or not or what tape will be placed on him.

The recommendations of the "Consolidated Standards of Reporting Trials" (CONSORT) will be followed. All participants will receive a participant information sheet and sign informed consent. Patients aged 18 to 65 years with low back pain will be recruited from different private clinics in the city of Valencia, Spain.

The hypothesis is that when Magnetic Tape® comes into contact with electromagnetic fields such as those generated by living beings, due to the movement of electrical charges (ions), as defined by Ampere's Law, the domains of the tape are oriented or aligned in parallel with the external magnetic field creating a magnetic flux with a north pole and a south pole. This generated field in turn produces a magnetic induction proportional to the variation of the magnetic flux, as defined by the Faraday Law.

This electric potential produces a redistribution of the electric charge (ions) generating a magnetic field due to the orientation of the tape domains, then exerting a force on the moving charges within the electrolyte.

Physiological, Lorentz's Law, regulating Magnetic Tape® aberrant electromagnetic fields.

The protocol for data collection will be as follows:

After signing the informed consent and data protection, the groups with low back pain will be formed that will receive the application of both Magnetic Tape® and the intervention of a placebo tape. To avoid that the order of the intervention influences the results of the study, the subjects will be randomized into two different groups, Group A and Group B. Group A will receive Magnetic tape® and Group B will do the opposite.

To standardize the location of the tape application, the patient will be placed in the prone position and the L4 spinous processes will be identified by marking them with a pen. Once L4 is located at the level of the iliac crests, the therapist will palpate the next spinous process down to the level of L5, and then it will be marked. The tape will be applied transversely covering the paravertebral skin at both levels.

Afte this protocol ultrasound will be applied, evaluating the characteristics of blood flow by means of ultrasound in the common femoral artery using pulsed power doppler. An Alpinion ECube 12 ultrsound machine with a L3-12H linear probe with a 64 mm footprint will be used. The variables of Peak systolic PS velocity in (cm/s), peak diastolic velocity (DF) in (cm/s), the difference between distolic an systolic (S/D), the pulsatility index (PI), the resistance index (IR) and the artery diameter in (cm) will be taken.

To assess pressure pain in the spinous processes, a Wagner Force Dial - FDK 20 algometer with a circular contact surface of 1 cm2 will be used. The sensation of perceived pain will be performed on the paravertebral skin of each level using the pinch technique and assessing it with the VAS scale. Both the algometer and pinch measurements will be repeated twice at each level leaving at least 1 minute between measurements.

During the pain measurement phase, each participant will be in the prone position where assessments will be made from L1 to S4. Afterwards, they will be placed in a supine position and for three minutes to adjust to the room environment and relax, the ultrasound measurements were taken. Subsequently, a tape will be placed and the perceived pain, pressure pain and vascular parameters will be measured again.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be subjects with low back pain aged 18-65 years residing in Valencia who wish to participate in the study.

Exclusion Criteria:

* not meeting the age requirement, having conditions that would be a contraindication to placing an adhesive bandage on the skin such as allergies, also being pregnant, having a pacemaker or people who have any contraindication of electromagnetic fields, neurological diseases or taking any medication that may interact with magnetic fields.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
peak systolic velocity (PSV) | 1 minute
  maximum systolic velocity of the femoral artery in (cm / s)
peak diastolic velocity (PDV) | 1 minute
  femoral artery peak diastolic velocity in (cm / s)
difference between systolic and diastolic (S / D) | 1 minute
  difference between systolic and diastolic in the femoral artery
pulsatility index (PI) | 1 minute
  assesses the peripheral resistance of blood vessels
resistance index (RI) | 1 minute
  reflects resistance to arterial flow
diameter | 1 minute
  diameter of each artery

SECONDARY OUTCOMES:
Algometria | 2 minutes
  referred pain when pressing on the lumbar vertebral processes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Francisco Selva, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No